CLINICAL TRIAL: NCT03992820
Title: The Efficacy of Transcutaneous Electrical Nerve Stimulation Versus Local Anaesthetic Cream in Alleviating the Pain of Local Anaesthetic Injections in Adults - A Randomised Controlled Trial
Brief Title: Transcutaneous Electrical Nerve Stimulation for Local Anaesthesia
Acronym: TENS-LA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped early due to COVID19 restrictions
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 113691
Record Dates: First submitted 2019-04-26; First posted 2019-06-20 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Donor Site Complication; Skin Graft
Keywords: TENS; local anaesthetic cream; skin graft donor site
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: After obtaining informed consent patients will be randomised to two groups using codes generated by web-based randomisation system- Research Randomizer. This is a free resource for researchers.
  The website is http://www.randomizer.org The numbers generated will be placed in separate sealed envelopes by the department secretary and made available to the investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TENS arm (trial arm) (Experimental): The trial group will have the TENS (transcutaneous electrical nerve stimulator) to the area planned for injection for at least 30 minutes before injection of the local anaesthetic solution.
  Interventions: Device: TENS machine
- EMLA arm (Control arm) (Other): The control group will have EMLA (Eutatic mixture of local anaesthetic) applied on the site planned for local anaesthetic injection and after 1 hour, will be removed and immediately injected with the same anaesthetic solution.
  Interventions: Combination Product: EMLA cream

INTERVENTIONS:
Device: TENS machine — The trial group will have the TENS to the area planned for injection for at least 30 minutes before injection of the local anaesthetic solution.
  Pain perception will be evaluated using two Numeric Pain Rating Scales in the study and control groups- one to assess the pain of needle penetration and the second to assess the pain of local infiltration.
  Arms: TENS arm (trial arm)
Combination Product: EMLA cream — The control group will have EMLA applied on the site planned for local anaesthetic injection and after 1 hour, will be removed and immediately injected with the same anaesthetic solution (this is already a procedure practised by many of the surgeons).
  Pain perception will be evaluated using two Numeric Pain Rating Scales in the study and control groups- one to assess the pain of needle penetration and the second to assess the pain of local infiltration.
  Arms: EMLA arm (Control arm)

SUMMARY:
TENS-LA trial is a randomised control trial to assess the possible efficacy of Transcutaneous Electrical Nerve Stimulation (TENS) on eliminating or reducing the pain of local anaesthetic injection for minor surgical procedures. Comparison is done with a mixture of local anaesthetic cream (EMLA) which is used at times for the same purpose. Though local procedures are carried out in various parts of the body, this trial will be conducted specifically on patients undergoing a split skin graft harvest from the thigh. Patients who meet the eligibility criteria and are willing to participate will be randomised to receive either TENS or EMLA.

Results will be analysed based on the pain score records at the end of the trial

DETAILED DESCRIPTION:
Patients undergoing a split skin graft harvest will be selected from theatre lists and will be given complete information regarding the nature of trial, possible complications, risks and advantages by sending them a Patient Information Sheet at least a week prior to the procedure when they are send an appointment. On the day of procedure, either the Chief Investigator or one of the other two Investigators will see the patient in the Theatre Arrivals Area and have a full discussion on the details of the trial and will answer all their questions. Patients willing to take part and are within the inclusion criteria and does not have any of the exclusion criteria will be randomised to either the study group or the control group after obtaining informed consent.

The trial group will have the TENS to the area planned for injection for 30 minutes before injection of the local anaesthetic (a combination of 0.25% levobupivacaine and 1% lignocaine with 1/200,000 adrenaline). The control group will have EMLA applied on the site planned for local anaesthetic injection and after 1 hour , will be removed and immediately injected with the same anaesthetic solution (this is already a procedure practised by some of the surgeons).

Pain perception will be evaluated using two Numeric Pain Rating Scales in the study and control groups- one to assess the pain of needle penetration and the second to assess the pain of local infiltration. The Numeric pain scale is filled in by the doctor as indicated by the patient. Pulse rate and Blood Pressure monitoring will be carried out as an objective measurement of response to pain (these are routinely recorded when patient is in the theater for a procedure). Patient involvement in the study ends at this point.

Analysis of the outcome will be done at the end of the trial period.

ELIGIBILITY:
Both interventions will be carried out in adult patients. For the purpose of standardisation and avoiding the variations from different sites in the body, and different surgical procedures, the site will be the thigh in both groups which is the donor site for a split skin graft.

Inclusion criteria:

• Adult patients aged 18 to 90 years undergoing a split skin graft harvest under local anaesthesia

Exclusion criteria:

* Patients below 18 and above 90 years of age
* Patients with dementia or other mental abnormalities causing incapacity.
* Pregnant ladies
* Patients with pace maker or ICD
* Patients with history of epilepsy or aneurysm
* Patients with undiagnosed skin or pain conditions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
The primary outcome is pain of local anaesthetic injection after application of TENS or LA cream as measured by two Numeric Pain Rating Scale | 10 minutes
  Pain perception will be evaluated using two Numeric Pain Rating Scales in the study and control groups. One scale will assess the pain caused by needle piercing the skin and the second will do so for the pain caused by infiltration of local anaesthetic agent.
  The scale used is "Numeric Pain rating scale" which shows a transverse line with values from 0 to 10 from left to right where 0 indicates no pain and 10 worst possible pain. The middle, which is 5 indicates moderate pain. Outcome of the intervention is better towards the left indicating less pain and worse towards the right indicating more pain.
  No sub scales are used.

SECONDARY OUTCOMES:
Changes in blood pressure in response to injection of local anaesthetic | 10 minutes
  Blood Pressure (BP) monitoring will be carried out as an objective measurement of response to pain. The unit of measurement is mm of Hg (millimetres of Mercury). This measurement is to assess if there is a rise in BP in response to the local anaesthetic injection after application of either TENS or EMLA and if present, to what extent. The changes will be analysed with respect to the baseline BP recording of the patient.
Changes in heart rate in response to injection of local anaesthetic | 10 minutes
  Heart rate (HR) monitoring will be carried out as an objective measurement of response to pain. The unit of measurement is number per minute. This measurement is to assess if there is a rise in HR in response to the local anaesthetic injection after application of either TENS or EMLA and if present, to what extent. The changes will be analysed with respect to the baseline HR recording of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Rajshree Jayarajan, Principal Investigator — University Hospitals, Leicester
Locations (1):
- University Hospitals of Leicester, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kasat V, Gupta A, Ladda R, Kathariya M, Saluja H, Farooqui AA. Transcutaneous electric nerve stimulation (TENS) in dentistry- A review. J Clin Exp Dent. 2014 Dec 1;6(5):e562-8. doi: 10.4317/jced.51586. eCollection 2014 Dec. PMID 25674327
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Mendell LM. Constructing and deconstructing the gate theory of pain. Pain. 2014 Feb;155(2):210-216. doi: 10.1016/j.pain.2013.12.010. Epub 2013 Dec 12. PMID 24334188
- [Background] Sluka KA, Deacon M, Stibal A, Strissel S, Terpstra A. Spinal blockade of opioid receptors prevents the analgesia produced by TENS in arthritic rats. J Pharmacol Exp Ther. 1999 May;289(2):840-6. PMID 10215661
- [Background] Kalra A, Urban MO, Sluka KA. Blockade of opioid receptors in rostral ventral medulla prevents antihyperalgesia produced by transcutaneous electrical nerve stimulation (TENS). J Pharmacol Exp Ther. 2001 Jul;298(1):257-63. PMID 11408550
- [Background] Wall PD, Sweet WH. Temporary abolition of pain in man. Science. 1967 Jan 6;155(3758):108-9. doi: 10.1126/science.155.3758.108. PMID 6015561
- [Background] Sluka KA, Bjordal JM, Marchand S, Rakel BA. What makes transcutaneous electrical nerve stimulation work? Making sense of the mixed results in the clinical literature. Phys Ther. 2013 Oct;93(10):1397-402. doi: 10.2522/ptj.20120281. Epub 2013 May 2. PMID 23641031
- [Background] Bjordal JM, Johnson MI, Ljunggreen AE. Transcutaneous electrical nerve stimulation (TENS) can reduce postoperative analgesic consumption. A meta-analysis with assessment of optimal treatment parameters for postoperative pain. Eur J Pain. 2003;7(2):181-8. doi: 10.1016/S1090-3801(02)00098-8. PMID 12600800
- [Background] Varadharaja M, Udhya J, Srinivasan I, Sivakumar JS, Karthik RS, Manivanan M. Comparative clinical evaluation of transcutaneous electrical nerve stimulator over conventional local anesthesia in children seeking dental procedures: A clinical study. J Pharm Bioallied Sci. 2014 Jul;6(Suppl 1):S113-7. doi: 10.4103/0975-7406.137407. PMID 25210350
- [Background] teDuits E, Goepferd S, Donly K, Pinkham J, Jakobsen J. The effectiveness of electronic dental anesthesia in children. Pediatr Dent. 1993 May-Jun;15(3):191-6. PMID 8378157
- [Background] 11. Choudhari SR, Parikrama SJ, Gaurav VK et al. Efficacy of transcutaneous electronic nerve stimulation in alleviating pain during inferior alveolar nerve block injections in pediatric dentistry. International Journal of Pedodontic Rehabilitation. 2017;2(2): 69-72
- [Background] Meechan JG, Gowans AJ, Welbury RR. The use of patient-controlled transcutaneous electronic nerve stimulation (TENS) to decrease the discomfort of regional anaesthesia in dentistry: a randomised controlled clinical trial. J Dent. 1998 Jul-Aug;26(5-6):417-20. doi: 10.1016/s0300-5712(97)00062-6. PMID 9699431
- [Background] Dhindsa A, Pandit IK, Srivastava N, Gugnani N. Comparative evaluation of the effectiveness of electronic dental anesthesia with 2% lignocaine in various minor pediatric dental procedures: A clinical study. Contemp Clin Dent. 2011 Jan;2(1):27-30. doi: 10.4103/0976-237X.79305. PMID 22114450
- [Background] Burri H, Piguet V. UninTENSional pacemaker interactions with transcutaneous electrical nerve stimulation. Europace. 2009 Mar;11(3):283-4. doi: 10.1093/europace/eup008. No abstract available. PMID 19240107
- [Background] Keskin EA, Onur O, Keskin HL, Gumus II, Kafali H, Turhan N. Transcutaneous electrical nerve stimulation improves low back pain during pregnancy. Gynecol Obstet Invest. 2012;74(1):76-83. doi: 10.1159/000337720. Epub 2012 Jun 21. PMID 22722614

DOCUMENTS (2):
  • Study Protocol (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT03992820/Prot_000.pdf
  • Informed Consent Form (2019-02-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT03992820/ICF_001.pdf